CLINICAL TRIAL: NCT01374048
Title: Are Intracranial Pressure Waves Measurable Through Lumbar Puncture?
Brief Title: Intracranial Pressure Waves Via Lumbar Puncture
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Anders Behrens MD, Department of Clinical Neuroscience
Other Study IDs: 97-88
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Idiopathic Normal Pressure Hydrocephalus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients are subjected to simultaneous intracranial and lumbar puncture pressure measurements. This study focus on intracranial pulse amplitude. Hypothesis: Intracranial pressure amplitude is reflected by lumbar puncture pressure amplitude.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Idiopathic Normal Pressure Hydrocephalus

Exclusion Criteria:

* Known cause of hydrocephalus

Ages: 55 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with idiopathic normal pressure hydrocephalus
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)